CLINICAL TRIAL: NCT06838130
Title: AI-Enhanced Analysis of Breast Density and Background Parenchymal Enhancement (BPE)
Status: Enrolling by invitation | Type: Observational
Sponsor: Link Campus University (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Graziella di Grezia, Principal Investigator, Link Campus University
Other Study IDs: T_6_2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Breast Parenchimal Enhancement; Artificial Intelligence (AI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patiens underwent CEM

SUMMARY:
This study expands upon previous research investigating the correlation between breast density, Background Parenchymal Enhancement (BPE), and age in contrast-enhanced mammography (CEM). By integrating Artificial Intelligence (AI) methodologies, including Artificial Neural Networks (ANNs) and deep learning models, the study aims to optimize the accuracy of predictions and validate prior findings obtained through multiple linear regression.

ELIGIBILITY:
Patients who underwent CEM, mammography, and ultrasound between May 2022 and June 2023.

Availability of BPE assessment, BI-RADS density classification, and age data.

Complete dataset available for statistical and AI-based analysis.

Exclusion Criteria:

Patients with prior breast cancer treatment that could alter BPE.

Incomplete imaging or missing classification data.

Contraindications to contrast-enhanced imaging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and older who underwent CEM for diagnostic or surveillance purposes.
  Patients with recorded BPE levels and BI-RADS breast density classification.
  Relational database containing structured data for correlation matrix analysis and AI model training.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between breast density, BPE, and age using AI-driven analysis. | Data analysis within 12 months of study completion.
  Evaluating whether AI models, including neural networks, can enhance prediction accuracy for BPE assessment compared to conventional multiple linear regression.

SECONDARY OUTCOMES:
AI-based optimization of breast density and BPE classification | Within 12 months of study completion
  Evaluating the performance of neural networks in predicting BPE levels across different breast density categories.
Comparative performance of multiple linear regression vs. AI models. | Within 12 months of study completion.
  Assessing the accuracy of traditional statistical methods versus ANN-based predictions in explaining variance in BPE values.
Mean Squared Error (MSE) and explained variance in predictive models | Within 12 months of study completion
  Analyzing the error rates and variance explained by different AI models compared to multiple linear regression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No